CLINICAL TRIAL: NCT00442559
Title: Korean Study of "Real-World" Montelukast Use in Mild Asthmatic Children With Concomitant Allergic Rhinitis
Brief Title: Montelukast in Mild Asthmatic Children With Allergic Rhinitis (0476-367)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0476-367; 2007_003
Record Dates: First submitted 2007-02-28; First posted 2007-03-02 (Estimated); Results first posted 2008-11-18 (Estimated); Last update posted 2024-05-13 (Actual); Status verified 2022-01

CONDITIONS: Asthma; Allergic Rhinitis
MeSH Terms: conditions — Asthma; Rhinitis, Allergic | interventions — montelukast

ARMS (2):
- Montelukast (Experimental): Participants were treated for 12 months after randomization: Participants 2 to 5 years of age took one 4 mg chewable tablet and 6 to 14 years of age took one 5 mg chewable tablet daily in the evening. If participants had exacerbated from mild to moderate within 12 weeks, inhaled corticosteroids (ICS) was added to Montelukast and ICS, respectively and those participants were excluded in the efficacy evaluation at 12 weeks.
  Interventions: Drug: montelukast sodium
- Inhaled Corticosteroids (ICS) (Active Comparator): Participants were treated for 12 months after randomization: Each participant's physician selected the ICS agent, dose, and regimen. If participants had exacerbated from mild to moderate within 12 weeks, ICS was added to Montelukast and ICS, respectively and those participants were excluded in the efficacy evaluation at 12 weeks.
  Interventions: Drug: inhaled corticosteroid

INTERVENTIONS:
Drug: montelukast sodium — Montelukast 4/5 mg tablet (oral chewable), once daily, 12 weeks to up to 12 months
  Other Names: Singulair, MK0476
  Arms: Montelukast
Drug: inhaled corticosteroid — Inhaled corticosteroid solution, 1-4 puffs daily, 12 weeks to up to 12 months
  Arms: Inhaled Corticosteroids (ICS)

SUMMARY:
The purpose of this study is to assess real-world effectiveness of montelukast in children (2 to 14 years) with asthma and allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Between 2 and 14 years old
* Diagnosed with asthma, classified as mild persistent asthma according to Global Initiative Asthma Guidelines (GINA)
* Diagnosed with comorbid allergic rhinitis

Exclusion Criteria:

* Patients with suspected sinus infection
* Prior treatment with high dose inhaled corticosteroid requiring a dose higher than beclomethasone dipropionate 400 ug per day, or equivalent, other medications used in severe cases

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 191 (Actual)
Dates: Start 2005-01; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Conducted at 5 sites in Korea, Jan2005~ Oct2007 in pediatric participants with comorbid mild asthma and allergic rhinitis. Participant's caregiver understands the study procedures and agrees to participate, signing the informed consent form.
Pre-assignment Details: Up to 1 week for wash-out - prior to baseline randomization.
Period: Overall Study
Arm/Group | Montelukast | Inhaled Corticosteroids (ICS)
Started | 100 | 91
12 Weeks After Randomization | 68 (12 weeks after randomization was pre-specified as the time point for analysis) | 60 (12 weeks after randomization was pre-specified as the time point for analysis)
Completed | 66 (12 weeks after randomization was pre-specified as the time point for analysis) | 56 (12 weeks after randomization was pre-specified as the time point for analysis)
Not Completed | 34 | 35
Not completed — Lost to Follow-up | 32 | 34
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Montelukast | Inhaled Corticosteroids (ICS) | Total
Number analyzed (Participants) | 24 | 29 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] — The primary efficacy parameter was a mean change from baseline to treatment for daytime asthma symptom score. Therefore 138 participants who didn't have a daytime asthma symptom score from the participant diary were not included.
  years | 5.4 (3.0) | 6.1 (2.6) | 5.8 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants] — The primary efficacy parameter was a mean change from baseline to treatment for daytime asthma symptom score. Therefore 138 participants who didn't have a daytime asthma symptom score from the participant diary were not included.
  Participants
    Female | 5 | 9 | 14
    Male | 19 | 20 | 39
Allergic rhinitis [Number; unit: participants] — Based on GINA guidelines. The primary efficacy parameter was a mean change from baseline to treatment for daytime asthma symptom score. Therefore 138 participants who didn't have a daytime asthma symptom score from the participant diary were not included.
  participants
    Mild-intermittent | 14 | 17 | 31
    Mild-persistent | 10 | 12 | 22
Type of allergic rhinitis [Number; unit: Participants] — The primary efficacy parameter was a mean change from baseline to treatment for daytime asthma symptom score. Therefore 138 participants who didn't have a daytime asthma symptom score from the participant diary were not included.
  Participants
    Seasonal | 13 | 15 | 28
    Perennial | 11 | 14 | 25
Daily allergic rhinitis symptom score [Mean (Standard Deviation); unit: Units on scale] — The score is an ordinal scale from 0 (no symptoms) to 3 (most symptoms). 24 participants with baseline scores were included in the Montelukast group and 28 participants with baseline scores were included in the ICS group.
  Units on scale | 0.45 (0.35) | 0.31 (0.34) | 0.37 (0.35)
Daytime asthma symptom score [Mean (Standard Deviation); unit: Units on scale] — The score is an ordinal scale from 0 (no symptoms) to 5 (most symptoms). The primary efficacy parameter was a mean change from baseline to treatment for daytime asthma symptom score. Therefore 138 participants who didn't have a daytime asthma symptom score from the participant diary were not included.
  Units on scale | 0.32 (0.42) | 0.29 (0.40) | 0.30 (0.40)
Duration of allergic rhinitis [Mean (Standard Deviation); unit: Years] — 24 participants were included in the Montelukast group and 28 participants were included in the ICS group.
  Years | 0.4 (0.6) | 0.8 (1) | 0.6 (0.9)
Duration of asthma [Mean (Standard Deviation); unit: Years] — The primary efficacy parameter was a mean change from baseline to treatment for daytime asthma symptom score. Therefore 138 participants who didn't have a daytime asthma symptom score from the participant diary were not included.
  Years | 0.6 (0.7) | 1.1 (1.2) | 0.9 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline for Daytime Asthma Symptom Score
Description: The score is an ordinal scale from 0 (no symptoms) to 5 (most symptoms). The change was calculated as the score at 12 weeks minus the score at baseline. Thus, a negative value for change from baseline indicates a favorable outcome.
Time Frame: Baseline and Week 12
Population: The primary efficacy parameter was a mean change from baseline to treatment for daytime asthma symptom score. Therefore 138 participants who didn't have a daytime asthma symptom score from the participant diary were not included.
Measure: Mean (Standard Deviation); unit: Units on scale
Groups:
- Daytime Asthma Symptom Score at Baseline - Montelukast; Daytime Asthma Symptom Score at 12 Weeks - Montelukast; Daytime Asthma Symptom Score at Baseline - ICS; Daytime Asthma Symptom Score at 12 Weeks - ICS: Participants received study drug and had efficacy measurements both at baseline and during the treatment period. If participants had exacerbated from mild to moderate within 12 weeks, inhaled corticosteroids (ICS) was added to Montelukast and ICS, respectively and those participants were excluded in the efficacy evaluation at 12 weeks.
Arm/Group | Daytime Asthma Symptom Score at Baseline - Montelukast | Daytime Asthma Symptom Score at 12 Weeks - Montelukast | Daytime Asthma Symptom Score at Baseline - ICS | Daytime Asthma Symptom Score at 12 Weeks - ICS
Number analyzed (Participants) | 24 | 24 | 29 | 29
Units on scale | 0.32 (0.42) [-0.29 to -0.03] | 0.16 (0.35) [-0.30 to -0.02] | 0.29 (0.4) | 0.13 (0.27)
Statistical Analysis 1: Comparison: Daytime Asthma Symptom Score at Baseline - Montelukast vs Daytime Asthma Symptom Score at 12 Weeks - Montelukast; Change from BL to Week 12 - Montelukast. The difference in mean change from baseline to 12 weeks in daytime asthma symptom score was tested by paired t-test (H0: difference =0) for the Montelukast treatment group. Subjects in this analysis: N=24 subjects for the within arm (single arm) comparison between BL and Week 12 scores; Test type: Superiority or Other; p = 0.015, t-test, 2 sided; Mean Difference (Final Values) = -0.16, 95% CI 2-sided [-0.29 to -0.03]
Statistical Analysis 2: Comparison: Daytime Asthma Symptom Score at Baseline - ICS vs Daytime Asthma Symptom Score at 12 Weeks - ICS; Change from BL to Week 12 - ICS. The difference in mean change from baseline to 12 weeks in daytime asthma symptom score was tested by paired t-test (H0: difference =0) for the ICS treatment group. Subjects in this analysis: N=29 subjects for the within arm (single arm) comparison between BL and Week 12 scores; Test type: Superiority or Other; p = 0.027, t-test, 2 sided; Mean Difference (Final Values) = -0.16, 95% CI 2-sided [-0.3 to -0.02]

2. Secondary Outcome: Change From Baseline for Daily Allergic Rhinitis Symptom Score
Description: The score is an ordinal scale from 0 (no symptoms) to 3 (most symptoms). The change was calculated as the score at 12 weeks minus the score at baseline. Thus, a negative value for change from baseline indicates a favorable outcome.
Time Frame: Baseline and Week 12
Population: The secondary efficacy parameter was a mean change from baseline to treatment for daily allergic rhinitis symptom score. Therefore 139 participants who didn't have a daily allergic rhinitis symptom score from the participant diary were not included.
Measure: Mean (Standard Deviation); unit: Units on scale
Groups:
- Daily Allergic Rhinitis Symptom Score at Baseline- Montelukast; Daily Allergic Rhinitis Symptom Score at 12 Weeks- Montelukast; Daily Allergic Rhinitis Symptom Score at Baseline - ICS; Daily Allergic Rhinitis Symptom Score 12 Weeks - ICS: Participants received study drug and had efficacy measurements both at baseline and during the treatment period. If participants had exacerbated from mild to moderate within 12 weeks, inhaled corticosteroids (ICS) was added to Montelukast and ICS, respectively and those participants were excluded in the efficacy evaluation at 12 weeks.
Arm/Group | Daily Allergic Rhinitis Symptom Score at Baseline- Montelukast | Daily Allergic Rhinitis Symptom Score at 12 Weeks- Montelukast | Daily Allergic Rhinitis Symptom Score at Baseline - ICS | Daily Allergic Rhinitis Symptom Score 12 Weeks - ICS
Number analyzed (Participants) | 24 | 24 | 28 | 28
Units on scale | 0.45 (0.35) [-0.36 to -0.07] | 0.23 (0.26) [-0.24 to -0.01] | 0.31 (0.34) | 0.19 (0.26)
Statistical Analysis 1: Comparison: Daily Allergic Rhinitis Symptom Score at Baseline- Montelukast vs Daily Allergic Rhinitis Symptom Score at 12 Weeks- Montelukast; Change from BL to Week 12 - Montelukast. The difference in mean change from baseline to 12 weeks in daily allergic rhinitis symptom score was tested by paired t-test (H0: difference =0) for the Montelukast treatment group. Subjects in this analysis: N=24 subjects for the within arm (single arm) comparison between BL and Week 12 scores; Test type: Superiority or Other; p = 0.006, t-test, 2 sided; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-0.36 to -0.07]
Statistical Analysis 2: Comparison: Daily Allergic Rhinitis Symptom Score at Baseline - ICS vs Daily Allergic Rhinitis Symptom Score 12 Weeks - ICS; Change from BL to Week 12 - ICS. The difference in mean change from baseline to 12 weeks in daily allergic rhinitis symptom score was tested by paired t-test (H0: difference =0) for the ICS treatment group. Subjects in this analysis: N=28 subjects for the within arm (single arm) comparison between BL and Week 12 scores; Test type: Superiority or Other; p = 0.032, t-test, 2 sided; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-0.24 to -0.01]

ADVERSE EVENTS:
Time Frame: Up to 12 months
Arm/Group | Montelukast | Inhaled Corticosteroids (ICS)
Serious Adverse Events (participants affected / at risk) | 4/100 | 3/91
Other Adverse Events (participants affected / at risk) | 83/100 | 70/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Montelukast (N=100) | Inhaled Corticosteroids (ICS) (N=91)
VOMITING (Gastrointestinal disorders) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 0 (0) | 1 (1)
CHRONIC SINUSITIS (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 1 (1) | 1 (1)
HEADACHE (Nervous system disorders) | 0 (0) | 1 (1)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Montelukast (N=100) | Inhaled Corticosteroids (ICS) (N=91)
VOMITING (Gastrointestinal disorders) | 6 (6) | 7 (7)
PYREXIA (General disorders) | 31 (41) | 24 (34)
NASOPHARYNGITIS (Infections and infestations) | 6 (6) | 2 (2)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 9 (9) | 7 (10)
HEADACHE (Nervous system disorders) | 9 (9) | 10 (11)
COUGH (Respiratory, thoracic and mediastinal disorders) | 56 (88) | 47 (92)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 7 (10) | 5 (6)
NASAL DISCOMFORT (Respiratory, thoracic and mediastinal disorders) | 15 (21) | 8 (9)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 8 (10)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 12 (17)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 27 (36) | 21 (30)
SNEEZING (Respiratory, thoracic and mediastinal disorders) | 21 (29) | 18 (26)
UPPER AIRWAY OBSTRUCTION (Respiratory, thoracic and mediastinal disorders) | 30 (42) | 30 (43)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 13 (15)

LIMITATIONS AND CAVEATS:
This was an open-label study. Only 53 patients had diary information with daytime asthma symptom score - thus, 138 cases were dropped from analysis due to lack of daytime asthma symptom score.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.